CLINICAL TRIAL: NCT06368024
Title: Establishment of Delphi-MD Safety Performance and Reliability
Status: Completed | Type: Observational
Sponsor: QuantalX Neuroscience (Industry)
Responsible Party: Sponsor
Other Study IDs: CL-12-600
Record Dates: First submitted 2023-11-26; First posted 2024-04-16 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Neurologic Disorder; Healthy
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is a retrospective analysis study of data collected with a diagnostic medical device — Transcranial Magnetic stimulation and Electroencephalogram

SUMMARY:
A retrospective analysis of collected datasets. In this study we aim to establish Delphi-MD's safety and performance reliability for assessment and monitoring of Transcranial Magnetic Stimulation (TMS) Evoked Potentials (TEPs) as neurophysiological measurements.

DETAILED DESCRIPTION:
A retrospective analysis of collected datasets. In this study we aim to establish Delphi-MD's safety and reliability for assessment and monitoring of TEP's as neurophysiological measurements.

Safety:

Upper limit of the 95% CI of the device related serious adverse event (SAE) rate is less than or equal to 3.6%

Performance:

Demonstrate differentiation of relevant clinical groups

Reliability:

An acceptable mean Interclass correlation (ICC) statistic (six stimulation) is at least 0.6 Additionally, the within subject variability should be lower than the between subject variability.

ELIGIBILITY:
Normal Population:

Inclusion Criteria:

1. Male and female subjects at the ages of 50-75.
2. With a technically-eligible EEG-TMS (Delphi-MD) evaluation recording performed

Exclusion Criteria:

1. Any neurodegenerative disease.
2. Neurological developmental disorder (e.g., Cerebral Palsy, Anoxic Brain Damage, Autism Spectrum Disorder).
3. Multiple Sclerosis (MS).
4. Major psychiatric disorders (e.g., Major Depressive Disorder, Generalized Anxiety Disorder, post traumatic stress disorder (PTSD), Bi-polar Disorder, Schizophrenia, Substance abuse),
5. Chronic central nervous system (CNS) pain disorders (Migraines, Fibromyalgia).
6. History of brain tumor, history of brain surgery or brain radiation damage.
7. Prior known epileptic episode.
8. Subjects with any metallic brain implant or fragments (such as shunt, pacemaker, clips, coils, bullet fragments, cochlear implants).
9. Subjects with any implanted devices activated or controlled by physiological signals and/or ferromagnetic or other magnetic sensitive metals implanted in the head or anywhere within 12 inches/30 cm from the stimulation coil.
10. Record of significant head trauma in the (e.g. loss of consciousness, altered consciousness, diagnosed evidence of contusion on brain imaging following trauma.
11. Current ongoing use of opioids, anti-psychotic, anti-epileptic, anti-depressant and Anxiolytics medications.
12. Intake of any other CNS directed medication such as sleeping pills 12 hours or less prior to the DELPHI evaluation.
13. Subjects that report drug abuse.
14. Pregnant or breastfeeding woman.

Clinical groups:

Inclusion criteria:

1. Men and women at the ages of >65
2. A clinical diagnosis of Dementia and/or Alzheimer's Disease, Lewy-Body Dementia (DLB), Parkinson's Disease, Normal Pressure Hydrocephalus (NPH) or stroke.

Exclusion criteria:

1. Subjects with any metallic brain implant or fragments (such as shunt, pacemaker, clips, coils, bullet fragments, cochlear implants).
2. Subjects with any implanted devices activated or controlled by physiological signals and/or ferromagnetic or other magnetic sensitive metals implanted in the head or anywhere within 12 inches/30 cm from the stimulation coil.
3. Record of significant head trauma in the (e.g. loss of consciousness, altered consciousness, diagnosed evidence of contusion on brain imaging following trauma.
4. Current ongoing use of opioids, anti-psychotic, or anti-epileptic medications.
5. Intake of any other CNS directed medication such as sleeping pills, SSRIs, Anxiolytics 12 hours or less prior to the DELPHI evaluation.
6. Subjects that report drug abuse.
7. Pregnant or breastfeeding woman.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and Female subjects at the ages of 50-75
Sampling Method: Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Cortical Excitability | baseline
  Amplitude of the TMS Evoked Response (TEP)- Mean amplitude deviation of the entire TEP time frame
Specific Peak Amplitudes | baseline
  N45,P60,N100,P180- Amplitudes at corresponding latencies
GMFP | baseline
  Global Mean Field Potential- It is a measure of the standard deviation of the potentials across all electrodes, reflecting the overall activity of the brain

CONTACTS AND LOCATIONS:
Locations (1):
- QuantalX Neuroscience Ltd., Kfar Saba, Center, Israel

IPD SHARING:
Plan to Share IPD: No